CLINICAL TRIAL: NCT02195401
Title: The Effects of a Clean Room Sleeping Environment on Elemental and Chemical Concentrations in Children and Adolescents With Autism Spectrum Disorders
Brief Title: The Effects of a Clean Room Sleeping Environment on Elemental and Chemical Concentrations in Children With Autism
Status: Completed | Type: Observational
Sponsor: The Children's Institute (Other)
Collaborators: Duquesne University (Other); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Dr. Scott Faber, Developmental Pediatrician, The Children's Institute
Other Study IDs: 09-131
Record Dates: First submitted 2014-07-16; First posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-07

CONDITIONS: Autism
Keywords: autism, cleanroom, immune dysregulation, toxins
MeSH Terms: conditions — Autistic Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Sleeping in a cleanroom: Each child and his or her parent slept in a cleanroom for two weeks. Within 24 hours pre and post this two week experience blood and hair samples were taken from the children and the parents filled out rating scales.
  Interventions: Other: Cleanroom

INTERVENTIONS:
Other: Cleanroom — Cleanroom with air the quality of the pre-industrial age

SUMMARY:
A child and their parent were asked to participate in a research project that sought to study whether sleeping in a very clean environment for 14 days improved the elimination of chemicals and metals from the child's body. The child had an approximately two hour evaluation to confirm his or her diagnosis of Autism or Pervasive Developmental Disorder. Not Otherwise Specified. When one of these diagnoses was confirmed the child was scheduled to spend 14 nights sleeping in a very clean environment in a specially created room at The Children's Institute.

Several hours prior to the first night the child slept in the clean room the child's mother, father, or guardian filled out behavioral rating scales about the child with the assistance of the study's research coordinator. The child also had approximately two tablespoons of blood drawn from an arm and a few inch sample of hair was taken from the back of the child's head. The child and a parent or guardian arrived at The Children's Institute about one half hour prior to the child's normal time of settling for bed for 14 consecutive nights. The child and a parent or guardian slept in the clean room, wearing the provided very clean clothes and sleeping on special mattresses and sheets each night for 14 consecutive nights. The child and parent were observed by a nurse through a window during the time in the clean room. The child and parent participated in regular daytime activities during these 14 days of the study. On the morning after the last night the child and a parent or guardian slept in the clean room a parent or guardian filled out behavioral rating scales with the help of the research coordinator. Approximately two tablespoons of blood were drawn from an arm and a few inch sample of hair was obtained from the back of the child's head, at The Children's Institute or at home.

DETAILED DESCRIPTION:
Autism spectrum disorders are characterized behaviorally by expressive language and social deficits, the performance of stereotypic and repetitive behavior patterns, and abnormal cognitive functioning. Children with autism spectrum disorders often do not have known anomalies seen on genetic testing. An emerging paradigm suggests that the majority of children with autism are displaying a pattern of genetic / environmental interaction that make them susceptible to difficulties with detoxification of the heavy metal and chemical environment. Children with autism demonstrate increased difficulty with the performance of methylation and sulfation required for the elimination of fat soluble chemicals from human tissues. These children also commonly display dysfunction of their metalloprotein systems necessary for the elimination of heavy metals such as mercury and arsenic from their bodies.

This study sought to provide 10 children with autism an opportunity to sleep in a clean room environment, a hospital room that was modified to remove nearly all traces of particulate matter, chemicals, and heavy metals, for a 2 week period while going about their normal activities during the day. In the clean room, the children slept on bedding and wore clothes that did not release any toxins. This room created a concentration gradient for chemical and heavy metal toxins that may have allowed these toxins to leave the children's bodies during their stays.

The children's parents filled out seven rating scales, including the Aberrant Behavior Checklist, immediately before and after the 2 week sleeping periods. The children had blood samples taken before and after the 2 week sleeping experiences that measured biomarkers of metalloprotein (heavy metal elimination) and immune functioning, such as the plasma zinc/serum copper ratio and T and B cell subsets. Red blood cell and hair concentrations of toxic heavy metals such as mercury, arsenic, and chromium 6, and red blood cell concentrations of chemicals implicated in contributing to human pathology, including polychlorinated biphenyls (PCBs), polybrominated diethyl ethers (PBDEs), and phthalates were determined before and after the sleeping experiences. These pre and post stay variables were statistically compared, and it was hypothesized that the children's red blood cell concentrations of toxins would be significantly reduced while their hair concentrations of toxins would be significantly increased after their sleeping experiences in the clean room, supporting the concept that the clean room promoted the release of heavy metals and chemicals from their bodies. This one year study was a proof of concept cohort study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of autism or Pervasive Developmental Disorder . Not Otherwise Specified
* Age 3-21
* Delayed verbal ability and limited academic skill sets that are advancing slowly with current programming

Exclusion Criteria:

* Children who are behaviorally severely dysregulated
* Children with other chronic medical conditions that require close monitoring
* Children with uncontrolled seizure disorder

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Ten children confirmed to have autism through ADOS
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in blood and hair elemental concentrations | Within one day pre and post 2 week experience of sleeping in the cleanroom

SECONDARY OUTCOMES:
Change of xenobiotic chemical concentrations | Within one day pre and post two week time the children sleep in the cleanroom

OTHER OUTCOMES:
Change of T and B cell subset results | Within one day pre and post the two week period the children sleep in the cleanroom

CONTACTS AND LOCATIONS:
Overall Officials: Scott Faber, MD, Principal Investigator — The Children's Institute; Skip Kingston, Ph.D., Principal Investigator — Duquesne University
Locations (1):
- The Children's Institute, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Faber S, Zinn GM, Boggess A, Fahrenholz T, Kern JC 2nd, Kingston HM. A cleanroom sleeping environment's impact on markers of oxidative stress, immune dysregulation, and behavior in children with autism spectrum disorders. BMC Complement Altern Med. 2015 Mar 19;15:71. doi: 10.1186/s12906-015-0564-0. PMID 25887094